CLINICAL TRIAL: NCT01592357
Title: The Effects of Tai Chi in Older Patients With Cardiovascular Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: McMaster University (Other)
Collaborators: Heart and Stroke Foundation of Ontario (Other); Hamilton Health Sciences Corporation (Other)
Responsible Party: Principal Investigator, Robert McKelvie, Professor of Medicine, Division of Cardiology, Medical Director, Heart Failure Program, HHS Medical Director, Cardiac Health and Rehabilitation Program, HHS, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NA7343
Record Dates: First submitted 2012-03-14; First posted 2012-05-07 (Estimated); Last update posted 2013-03-19 (Estimated); Status verified 2013-03

CONDITIONS: Cardiovascular Disease
Keywords: cardiac rehabilitation; gait speed; mind body exercise; tai chi; cardiac disease; frail elderly
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases | interventions — Aquatic Therapy; Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tai Chi (Experimental)
  Interventions: Behavioral: Tai Chi exercise
- Sham Exercise (Sham Comparator)
  Interventions: Behavioral: Sham Exercise

INTERVENTIONS:
Behavioral: Tai Chi exercise — A short and simple 8-forms Tai Chi routine will be used in this study. This routine has been previously standardized and field tested. Participants will be coached, by a certified Tai Chi instructor, in practicing the proper mechanics of executing each of the eight physical movements comprising the 8-forms of Tai Chi. A brief 5 minute period of walking calisthenics pertinent to Tai Chi movements, postures and diaphragmatic breathing will take place before training to warm up and after training to cool down. The Tai Chi training will be 2 times a week and the total exercise time, including warm-up and cool down, will be 50 minutes for each session. Over a period of 12 weeks, the participants will learn all 8-forms and continue practicing them for the final 12 weeks of the training period.
  Arms: Tai Chi
Behavioral: Sham Exercise — The sham exercise (control) group will be involved in low-intensity stretching exercises two times per week. These exercises will be designed as a "sham exercise" condition. A brief 5 minute period of walking will take place before the sham exercise to warm up and after the sham exercise to cool down. Sham exercise sessions will include stretching exercises of the neck, trunk and extremities. The total exercise time for the "sham exercise" group will be 50 minutes and participants will meet 2 times per week for a period of 24 weeks.
  Other Names: Control Group
  Arms: Sham Exercise

SUMMARY:
Cardiac exercise rehabilitation consists of walking and bicycling activities. As the population requiring rehabilitation is aging, other forms of exercise may be useful and better tolerated. Tai Chi has been used for centuries, is easy to perform even by more debilitated individuals, and promotes improvement in blood pressure, fitness, and relaxation. Tai Chi may be more beneficial for frail cardiac patients because it is especially suited for the unfit and elderly, and can be practiced anywhere. Further studies are required to assess this form of exercise in cardiac patients. The objective of this randomized controlled study is to compare the effects of Tai Chi to "sham exercise" training in 200 frail cardiac patients who have completed six months of cardiac rehabilitation and are 60 years of age or older. Participants will be randomized to Tai Chi or "sham exercise" training and have their gait speed, blood pressure, heart rate, exercise capacity, balance, quality of life and cognitive function assessed before and after 24 week of training.

DETAILED DESCRIPTION:
The role of exercise training is well established for cardiac patients to improve fitness and clinical outcomes. Many older cardiac patients even if they initially participate do not maintain regular exercise for a number of reasons. As the population ages there is a need to evaluate other forms of exercise training that may be used alone or in conjunction with standard approaches. Tai Chi is a potentially beneficial exercise for older cardiac patients because it is low-intensity exercise especially suited for unfit and elderly patients. There has been little rigorous evaluation, especially in the cardiac populations, of Tai Chi.

The main objective of this study is to assess the effects of Tai Chi compared to "sham exercise" in cardiac patients that have completed a program of cardiac rehabilitation. The investigators hope to show that six months of Tai Chi training compared to "sham exercise" (with all participants instructed to maintain their standard exercise program), will improve gait speed, exercise capacity, health related quality of life, cognitive function and balance.

This is a single blind randomized controlled trial of 200 cardiac patients, great than or equal to 60 years of age, who have completed six months of cardiac rehabilitation at the Hamilton Health Science Cardiac Health and Rehabilitation Centre. Participants will be randomized to receive either the short and simple 8-forms Tai Chi routine or "sham exercise". The participants in the study will train for a period of six months.

ELIGIBILITY:
Inclusion Criteria:

1. Walking Speed < or = 1.3 m/sec during the gait speed assessment.
2. Evidence of cardiovascular disease based on a diagnosis of previous myocardial infarction, angiographic findings of coronary artery disease, previous percutaneous coronary intervention, or previous coronary artery bypass graft surgery.
3. Local resident, with available transportation to the Cardiac Health and Rehabilitation Centre (CHRC) at the Hamilton Health Sciences General Division.
4. Ability to understand written and verbal instructions and provide written informed consent.
5. Stable cardiac medical therapy as demonstrated by no change in medication during the 3 months prior to randomization.
6. Previous completion of the 6 month Cardiac Rehabilitation program (including exercise training component) at the CHRC.

Exclusion Criteria:

1. New York Heart Association Functional class IV symptoms of shortness of breath or angina.
2. Development of angina or ST segment depression of > 1 mm during symptom limited exercise testing at < 80% of predicted maximum power output.
3. Development of dysrhythmias during exercise (> Lown grade 2).
4. Resting blood pressure greater than 160 mmHg systolic or 90 mmHg diastolic.
5. Abnormal blood pressure response to clinical exercise testing (decrease in systolic pressure below resting; decrease of > 20 mmHg in systolic pressure after the normal exercise increase; rise in diastolic blood pressure of > 15 mmHg; maximal systolic blood pressure in excess of 250 mmHg).
6. Maximum heart rate < 100 beats per minute in the absence of beta blocker therapy.
7. Respiratory limitation as assessed by pre-exercise pulmonary function testing (documented restrictive or obstructive lung disease; based on forced expired volume in 1 sec and/or vital capacity measurements < 70% of predicted).
8. Major orthopedic disability.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-11; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Gait speed following 6 months of Tai Chi or sham exercise training | 24 weeks
  Gait speed will be measured by having participants walk a 4 metre course at their usual speed. There will be a 1-metre start-up before starting the timing for the walk over 4 metres. Each participant will be timed for 2 walks and the faster of the 2 walks will be used in the analysis.

SECONDARY OUTCOMES:
Peak exercise oxygen uptake (VO2) | 24 weeks
  Peak VO2 will be measured while performing cycle ergometry exercise.
Resting heart rate | 24 weeks
  Resting heart rate will be measured prior to participant performing a cycle ergometry exercise test.
Blood pressure | 24 weeks
  Blood pressure will be measured prior to the participant performing a cycle ergometry exercise test.
Balance assessment | 24 weeks
  Balance will be measured using the functional reach assessment and the single leg stance assessment.
Health related quality of life (HRQOL) | 24 weeks
  The Medical Outcomes Short Form 36 will be used to measure HRQOL.
Cognitive function following 6 months of Tai Chi or sham exercise training | 24 weeks
  Cognitive function will be measured using the Montreal Cognitive Assessment (MoCA) questionnaire (Version 7.1).

CONTACTS AND LOCATIONS:
Overall Officials: Robert S McKelvie, MD, PhD, Principal Investigator — Hamilton Health Sciences Corporation; Heather M Arthur, PhD, Study Chair — McMaster University; George Heckman, MD, MSc, Study Chair — University of Waterloo; Noori Akhtar-Danesh, PhD, Study Chair — McMaster University; Maureen MacDonald, PhD, Study Chair — McMaster University
Locations (1):
- Cardiac Health & Rehabilitation Centre, Hamilton Health Sciences, Hamilton, Ontario, Canada